CLINICAL TRIAL: NCT06249971
Title: A Single-stage Bilayered Skin Reconstruction Using Glyaderm® as an Acellular Dermal Regeneration Template Results in Improved Scar Quality: an Intra-individual Randomized Controlled Trial
Brief Title: A Single-stage Bilayered Skin Reconstruction With Glyaderm®
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Research Foundation Flanders (Other)
Responsible Party: Principal Investigator, Phillip Blondeel, Professor Dr Stan Monstrey, University Hospital, Ghent
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B670201733327
Record Dates: First submitted 2024-01-18; First posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-01

CONDITIONS: Burns; Full Thickness Burn; Necrotizing Fascitis
MeSH Terms: conditions — Burns; Fasciitis, Necrotizing | interventions — Skin Transplantation

STUDY DESIGN:
Intervention Model Description: A prospective, randomized, controlled, intra-individual, single-blinded study in a mono-center setting
Who Masked: Participant
Masking Description: Randomization only known to the surgeon and burn care coordinators, not the patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Split thickness skin graft alone (Active Comparator): Intra-individual approach Patient has 2 comparable (near) full thickness skin defects or 1 (near) full thickness skin defect that can be divided into 2 comparable regions.
  Randomization: the defect randomized in this arm receives only a skin graft.
  Interventions: Procedure: Skin graft alone
- Split thickness skin graft + Glyaderm (Experimental): Intra-individual approach Patient has 2 comparable (near) full thickness skin defects or 1 (near) full thickness skin defect that can be divided into 2 comparable regions.
  Randomization: the defect randomized in this arm receives a skin graft combined with Glyaderm
  Interventions: Procedure: Dermal subsitute Glyaderm + skin graft

INTERVENTIONS:
Procedure: Dermal subsitute Glyaderm + skin graft — A human donor-derived dermal substitute will be implanted together with a skin graft
  Arms: Split thickness skin graft + Glyaderm
Procedure: Skin graft alone — Skin graft alone with no dermal substitute
  Arms: Split thickness skin graft alone

SUMMARY:
The study will explore the potential of utilizing Glyaderm® in a single-stage engrafting process, aiming for a more cost-effective approach. While the absence of the reticular dermal layer is a challenge associated with autologous split-thickness skin grafting (STSG), often leading to hypertrophic scars and contractures, various dermal substitutes with inconsistent results exist. Bilayered skin reconstruction using glycerolized acellular dermis (Glyaderm®) has shown promise in improving scar quality through a two-step procedure. However, unlike the typical two-step process required for most dermal substitutes, our investigation focuses on the cost-effective application of Glyaderm® in a single-stage engrafting. This approach, if successful, could offer advantages such as reduced costs, shorter hospitalization times, and lower infection rates-attributes preferred by many surgeons, especially when autografts are available.

DETAILED DESCRIPTION:
BACKGROUND. Patients suffering from severe burn injury are often confronted with life-threatening complications such as absence of the protective skin barrier which eventually lead to infections, sepsis and even death. The standard therapy for deep and full thickness burns consists of surgical debridement and coverage with autologous split thickness skin grafts (STSG) which normally results in a fast closure of the wounds contributing to an increased survival rate for burn victims. However, these thin skin grafts almost exclusively consist of epidermis only and due to the absence of most of the thicker dermal layer, which is crucial for the mechanical properties of the skin, the healing of these burn wounds inevitably results in hypertrophic and unaesthetic scar formation and contractures. Subsequently a long and difficult rehabilitation follows often with in the end poor aesthetic and functional long-term results and frequent psychological problems. Ideally, both skin layers (epidermis+dermis) should be reconstructed to improve the scar quality and therefore the quality of life after burns. As a consequence, dermal substitutes are necessary but the extremely high cost of all currently available dermal substitutes still is a major obstacle for its widespread application.

SCIENTIFIC APPROACH. At the burn center of the Ghent University Hospital a significant amount lot of research has been targeted towards the development of a dermal substitute based on glycerolized allogenic skin grafts (Glyaderm). The use of human skin for dermal substitutes is ideal because the natural 3D network of collagen and elastin fibers is already provided and can be preserved. In order to prevent rejection our research group, together with the Euro Tissue Bank (ETB), developed a method of decellularization with a low concentration of sodium hydroxide (NaOH). Previous publications from our research team have demonstrated the beneficial effects of Glyaderm compared to STSG-only application. Unfortunately, our initial protocol required an additional surgical procedure to allow for optimal ingrowth of the dermal substitute before the STSG could be applied. This increased not only the time to healing but also the costs involved. Within the last two years a pilot study has demonstrated that further optimization of the substitute and of the procedure resulted in a successful simultaneous application of Glyaderm and STSG. The scientific objective of this project is to obtain the necessary clinical evidence for this improved applicability of Glyaderm in deep burns or full thickness skin defects by providing a bilayered reconstruction of the skin with simultaneous application of this dermal substitute combined with a STSG in a one surgical procedure. The scientific approach will consist of performing a large prospective, controlled, randomized, intra-individual comparative clinical study, investigating simultaneous application of Glyaderm + STSG versus STSG alone in deep burns and other full thickness skin defects. Power calculation determined that a total of 75 patients must be included: both early outcome parameters (graft take, ingrowth, and time to healing) as well as late outcome measurements (scar characteristics, quality of life, histology) will be evaluated up to 12 months post burn.

UTILIZATION. A recent report of the Kennis Centrum/Centre d'Expertise (KCE) demonstrated that each year more than 2500 (severely) burned patients are admitted to a Belgian hospital or burn center with the majority of them requiring surgical therapy (ref). The utilization objective of this project is to make Glyaderm universally available for the treatment of patients with deep burns or other full thickness skin defects. This effective, low-cost and easy-to-use dermal substitute should facilitate the patient's rehabilitation by providing a more aesthetic scar formation with less functional impairment. The ultimate goal is an improved quality of life for the patient with a better reintegration of the burn victims into society. Our utilization strategy will focus on the actual application of the study results for the patient's well-being and an important role hereby is reserved for the Advisory Committee. For this purpose we have extended an already existing network of major stakeholders who all are committed to the clinical utilization process. Included in this group are representatives of: patients' self-help groups, the Belgian Burn Foundation, an inter-mutualistic committee, a representative from the RIZIV (national health care reimbursement organization), of health economics and from Belgian and Dutch tissue banks. If indeed the results of our clinical study demonstrate an improved aesthetic and functional outcome as well as a significant reduction in time to heal and operative costs, then this should eventually lead to a better reimbursement, even in the current era of budget restrictions. Implementation of Glyaderm as a readily-available and easy to use reconstructive tool into the existing armamentarium of the surgeon will be realized through workshops, training courses as well as presentation in national and international congresses.

The ultimate goal is to establish a universal application of this cost-effective dermal substitute in Flanders and due to the simplicity of the decellularization procedure also throughout Belgium and even worldwide. Glyaderm could be used on all aesthetically or functionally important places and even more so in children and in economically disadvantaged patients.

ELIGIBILITY:
Inclusion Criteria:

* All deep partial thickness and full-thickness burns as shown by laser Doppler imaging (LDI) and/or clinically evaluated by two plastic surgeons or a burn care coordinator
* Other full-thickness skin defects besides burns, e.g. necrotizing fasciitis, deglovements or phalloplasty donor sites after free flap harvest
* Possibility to follow the complete treatment schedule until final graft take and subsequently wound healing and participation in the follow-up schedule
* Informed consent has been obtained • Age between 18-80 years

Exclusion Criteria:

* All partial-thickness burns that can heal by conservative treatment confirmed by LDI • Not completing the treatment schedule or declining further follow-up • The patient has any condition(s) that seriously compromises the patient's ability to complete this study. • The patient has participated in another study utilizing an investigational drug within the previous 30 days • The patient has one or more medical condition(s) that, in the opinion of the investigator, would make the patient an inappropriate candidate for this study e.g. diabetes, renal or hepatic insufficiency, immune or neurologic disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Graft take | 7 days
  take of the skin graft 6 days post-surgery, expressed as a percentage
healing time | up to 1 month
  the time needed until the wound is at least 95% closed AND does not need a significant wound dressing. Expressed in days.
bacterial load | up to 1 month
  The bacterial load is the amount of bacteria that is present in the wound, assessed with a wound swab. The bacterial load is expressed on a semi-quantative scale -,+,++,+++

SECONDARY OUTCOMES:
scar hydration | 1 year
  the hydration state of the stratum corneum of the scar. Expressed in arbitrary units.
scar water evaporation | 1 year
  the evaporation of water at the level of the stratum corneum of the scar as measured by the Tewameter. Expressed in g/h/m²
scar elasticity | 1 year
  the elasticity of the scar as measured by the cutometer. Expressed in arbitrary units.
extracellular matrix formation | 1 year
  the organization of the extracellular matrix as assessed by light microscopy on a biopsy. Expressed on a numerical scale of 0-5 from not present to well organized.
scar color, erythema | 1 year
  The redness of the scar as measured by the mexameter. Expressed in arbitrary units.
scar color, pigmentation | 1 year
  amount of pigmentation present in the scar as measured by the mexameter. Expressed in arbitrary units.

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University Hospital, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
Share all data in scientific publication

REFERENCES:
- [Background] De Decker I, Hoeksema H, Verbelen J, De Coninck P, Speeckaert M, De Schepper S, Blondeel P, Pirayesh A, Monstrey S, Claes KEY. A single-stage bilayered skin reconstruction using Glyaderm(R) as an acellular dermal regeneration template results in improved scar quality: an intra-individual randomized controlled trial. Burns Trauma. 2023 May 2;11:tkad015. doi: 10.1093/burnst/tkad015. eCollection 2023. PMID 37143955